CLINICAL TRIAL: NCT05324072
Title: Prevalence and Risk Factors of Work Related Musculoskeletal Disorders Among Egyptian Anesthesiologists: a Cross-sectional Study.
Brief Title: Musculoskeletal Disorders Among Egyptian Anesthesiologists
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hosam eldeen Marie, MD, Sohag University
Other Study IDs: 314450
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — observational study

SUMMARY:
This cross-sectional online survey questionnaire based study for Prevalence and risk factors of work related musculoskeletal disorders among Egyptian anesthesiologists.

DETAILED DESCRIPTION:
This cross-sectional online survey questionnaire based study will be approved by medical ethical committee of Sohag faculty of medicine. Survey participants will be reassured that all data collected are for research purposes. Responses will be voluntary anonymous and have no identifying data. Egyptian anaesthesiologists will be invited through social media to participate in the survey.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian anesthesiologists on clinical practice

Exclusion Criteria:

-

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Egyptian anesthesiologists on practice inside or outside Egypt
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of work related musculoskeletal disorders among Egyptian anesthesiologists | April to September 2022

SECONDARY OUTCOMES:
Risk factors of work related musculoskeletal disorders among Egyptian anesthesiologists | April to September 2022

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa Mohammed, MD, Study Director — Sohag Faculty of medicine
Locations (1):
- Sohag faculty of medicine, Aswān, Please Select, Egypt

IPD SHARING:
Plan to Share IPD: Undecided